CLINICAL TRIAL: NCT07212413
Title: Postoperative Sensitivity in Class II Restorations: A Randomized Clinical Trial Comparing Snow-Plow and Resin Coating Techniques
Brief Title: Effect of Snow-plow Technique on the Postoperative Pain Following Direct Composite Restoration
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Alaa Al-Haddad, Assisstant profossor in restorative dentistry, University of Jordan
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2/5/1/200
Record Dates: First submitted 2025-09-30; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: Postoperative Tooth Sensitivity Following Class II Composite Restorations
Keywords: Postoperative sensitivity; Class II composite restoration; Snow-plow technique; Resin coating technique; Pain assessment

STUDY DESIGN:
Intervention Model Description: A randomized split-mouth clinical trial with two intervention arms (snow-plow and resin coating techniques) allocated to contralateral Class II cavities in the same patient. This crossover model minimizes inter-individual variability by enabling within-subject comparison under identical clinical conditions.
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor was blinded to the restorative technique used on each tooth. Telephone interviews were conducted using standardized scripts, and the interviewer was unaware of the allocation, referring to teeth by quadrant/side to minimize bias. The operator is not blinded due to the nature of the restorative procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Snow-plow technique (Experimental): Class II posterior cavities were restored using the snow-plow technique. After adhesive application, a thin layer of uncured flowable bulk-fill resin was placed on the gingival floor. A packable bulk-fill composite was then immediately inserted, displacing the flowable resin, and both were light-cured simultaneously. The occlusal anatomy was completed with packable composite, followed by finishing and polishing. Rubber-dam isolation and selective enamel etching with a universal adhesive were applied in all cases.
  Interventions: Procedure: Snow-plow restorative technique
- Resin coating technique (Experimental): Class II posterior cavities were restored using the resin coating technique following immediate dentin sealing. After adhesive application, a thin layer of flowable bulk-fill resin was applied and light-cured to create a stress-absorbing layer on the dentin surface. Packable bulk-fill composite was then used to restore the remaining cavity, followed by occlusal sculpting, finishing, and polishing. All procedures were performed under rubber-dam isolation with selective enamel etching and universal self-etch adhesive on dentin.
  Interventions: Procedure: Resin coating restorative technique

INTERVENTIONS:
Procedure: Snow-plow restorative technique — The snow-plow technique involves placing a thin layer of uncured flowable bulk-fill resin on the gingival floor of a Class II cavity, immediately followed by placement of a packable bulk-fill composite. Both materials are light-cured simultaneously, allowing the flowable resin to fill voids and improve marginal adaptation.
  Other Names: Snowplow technique
  Arms: Snow-plow technique
Procedure: Resin coating restorative technique — The resin coating technique involves applying and light-curing a thin layer of flowable bulk-fill resin after adhesive application to create a stress-absorbing layer on dentin (resin coating), followed by restoration with packable bulk-fill composite. This approach aims to protect the dentin, enhance bond stability, and reduce postoperative sensitivity
  Other Names: Resin coating; Immediate dentin sealing with flowable liner
  Arms: Resin coating technique

SUMMARY:
This study is designed to compare two modern techniques used to restore decayed back teeth with tooth-colored filling materials. Some patients experience temporary discomfort or sensitivity after these types of dental treatments. The purpose of this study is to learn whether one technique may help reduce this short-term sensitivity compared to the other.

Adults who need fillings on both sides of their mouth are invited to participate. Each patient will receive one filling using each technique, placed in different teeth during the same appointment. The procedures will be performed using standard clinical methods and materials.

After treatment, participants will be contacted by telephone to report any discomfort at several time points during the first week. The interviewer will not know which technique was used for each tooth to ensure unbiased reporting. This information will help dentists better understand how these techniques affect patients' comfort in the days following treatment.

DETAILED DESCRIPTION:
Postoperative tooth sensitivity is a common but often transient symptom following the placement of direct posterior resin composite restorations. Patients frequently report mild to moderate discomfort, particularly during the first few days after treatment, which can influence their perception of treatment success and overall satisfaction. While advances in adhesive dentistry and restorative materials have greatly improved clinical outcomes, postoperative sensitivity remains a relevant clinical concern.

This clinical trial is designed to compare two contemporary restorative techniques-the snow-plow technique and the resin coating technique following immediate dentin sealing-in terms of postoperative patient-reported pain during the first postoperative week. Both techniques aim to enhance marginal adaptation and reduce polymerization shrinkage stresses at the adhesive interface, thereby potentially minimizing pulpal irritation and postoperative discomfort.

Participants in this study are adult patients requiring Class II resin composite restorations on two comparable posterior teeth, typically located on opposite sides of the dental arch. Each participant will receive two restorations, one using the snow-plow technique and the other using the resin coating technique, in a split-mouth design. This approach allows each participant to serve as their own control, minimizing inter-patient variability and enabling a more reliable comparison between the two restorative strategies.

All procedures are performed under rubber dam isolation using standardized adhesive and restorative protocols to ensure clinical consistency. The snow-plow technique involves placing an uncured flowable bulk-fill resin on the cavity floor, immediately followed by the placement of a packable composite increment. Both materials are then light-cured simultaneously. This technique is intended to improve adaptation of the restorative material to cavity walls, displace voids, and reduce microleakage.

In the resin coating technique, immediate dentin sealing is performed following cavity preparation. A thin layer of flowable bulk-fill resin is then applied over the sealed dentin and light-cured before the placement of the final packable composite increment. This layer acts as a stress-absorbing liner, providing a flexible interface that may protect the pulp and reduce the transmission of shrinkage stresses during polymerization.

Operator calibration and adherence to standardized protocols are emphasized to ensure uniformity. All restorations are carried out by a single experienced clinician using the same materials, instruments, and curing devices to reduce variability related to operator technique.

Postoperative discomfort is assessed using a standardized visual analog scale (VAS) during structured telephone interviews conducted at baseline (before treatment), 24 hours, 72 hours, and one week postoperatively. Interviews are performed by an assessor who is blinded to the restorative technique used for each tooth to minimize reporting bias. Participants are specifically instructed to evaluate each treated tooth independently without making side-by-side comparisons.

This study does not involve any experimental drugs or non-standard clinical procedures. Both restorative techniques are widely accepted in routine clinical practice and use materials that are commercially available and approved for dental use. The primary objective is to evaluate the early postoperative pain experience associated with each technique, rather than to introduce a novel material or intervention.

The findings of this study will contribute to a better understanding of how restorative technique selection influences postoperative sensitivity, potentially informing evidence-based clinical decision-making in restorative dentistry. By comparing two established but mechanistically distinct approaches, this trial aims to provide clinically relevant information that may help dentists optimize patient comfort following posterior resin composite placement.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18-50 years.
* Systemically healthy individuals.
* Presence of two posterior teeth in different quadrants or contralateral sides of the same arch requiring Class II composite restorations.
* Teeth diagnosed with reversible pulpitis and vital pulps, confirmed clinically and radiographically.
* Teeth without previous restorations or carious lesions limited to dentin.
* Ability to provide informed consent and comply with study procedures and follow-up assessments.

Exclusion Criteria:

* Non-vital teeth, teeth with signs of irreversible pulpitis, periapical pathology, or extensive loss of tooth structure.
* Patients with systemic conditions or medications that may influence pain perception, healing, or sensitivity (e.g., chronic pain syndromes, analgesic use, immunosuppressive therapy), or very poor oral hygiene.
* Pregnant or breastfeeding women.
* Known allergy to dental materials used in the study.
* Inability to respond to follow-up calls or provide reliable pain assessments.
* Teeth with previous restorations, endodontic treatment, or cracks.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2025-01-12 (Actual); Primary Completion 2025-09-24 (Actual); Study Completion 2025-10-06 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain intensity after Class II composite restorations | Baseline, 24 hours, 72 hours, and 1 week after restorative treatment
  Postoperative pain intensity will be assessed using a 0-10 Visual Analog Scale (VAS) at baseline (before treatment), 24 hours, 72 hours, and 1 week following restorative procedures. Each treated tooth will be evaluated individually using structured telephone interviews conducted by a blinded examiner. VAS scores will be recorded and analyzed to compare pain trajectories between the snow-plow and resin coating restorative techniques.

CONTACTS AND LOCATIONS:
Overall Officials: Alaa Al-Haddad, PhD, Principal Investigator — University of Jordan
Locations (1):
- Univeristy of Jordan Hospital, Dental Department, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the results will be shared, including demographic data, intervention assignment, and all primary and secondary outcome measures. Data will be available to qualified researchers upon reasonable request following publication of the study results, in accordance with institutional and ethical guidelines. Supporting materials, such as the study protocol and statistical analysis plan, will also be provided.
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Background] Afifi SMH, Haridy MF, Farid MR. Evaluation of Post-Operative Sensitivity of Bulk Fill Resin Composite versus Nano Resin Composite: A Randomized Controlled Clinical Study. Open Access Maced J Med Sci. 2019 Jul 26;7(14):2335-2342. doi: 10.3889/oamjms.2019.656. eCollection 2019 Jul 30. PMID 31592052
- [Background] Lehmann A, Nijakowski K, Jankowski J, Donnermeyer D, Ramos JC, Drobac M, Martins JFB, Hatipoglu O, Omarova B, Javed MQ, Alharkan HM, Bekjanova O, Wyzga S, Alkhawas MAM, Kudenga R, Surdacka A. Clinical Difficulties Related to Direct Composite Restorations: A Multinational Survey. Int Dent J. 2025 Apr;75(2):797-806. doi: 10.1016/j.identj.2024.06.012. Epub 2024 Jul 23. PMID 39048490
- [Background] Tee R, Vach K, Schlueter N, Jacker-Guhr S, Luehrs AK. High C-Factor Cavities: How Do "Snowplow Technique", Adhesive Application Mode and Aging Influence the Microtensile Bond Strength to Dentin? J Adhes Dent. 2024 Jan 15;26:1-10. doi: 10.3290/j.jad.b4835909. PMID 38224111
- [Background] Putignano A, Tosco V, Monterubbianesi R, Vitiello F, Gatto ML, Furlani M, Giuliani A, Orsini G. Comparison of three different bulk-filling techniques for restoring class II cavities: muCT, SEM-EDS combined analyses for margins and internal fit assessments. J Mech Behav Biomed Mater. 2021 Dec;124:104812. doi: 10.1016/j.jmbbm.2021.104812. Epub 2021 Sep 3. PMID 34500356
- [Background] Tardem C, Albuquerque EG, Lopes LS, Marins SS, Calazans FS, Poubel LA, Barcelos R, Barceleiro MO. Clinical time and postoperative sensitivity after use of bulk-fill (syringe and capsule) vs. incremental filling composites: a randomized clinical trial. Braz Oral Res. 2019 Sep 16;33(0):e089. doi: 10.1590/1807-3107bor-2019.vol33.0089. PMID 31531552
- [Background] Miletic V, Komlenic V, Bajuk-Bogdanovic D, Stasic J, Petrovic V, Savic-Stankovic T. Preheating and "snow-plow" composite application technique affect double bond conversion but not bond strength to dentine. J Esthet Restor Dent. 2024 Jun;36(6):951-961. doi: 10.1111/jerd.13218. Epub 2024 Mar 18. PMID 38497672